CLINICAL TRIAL: NCT02259998
Title: An Open-labelled, Randomised, 2-way Crossover Study to Compare the Pharmacokinetics of Two Different Persantin® Sugar Coated Tablets 75 mg p.o. (Present and Proposed Formulation in France) q.i.d. for Three Days in Healthy Male Volunteers
Brief Title: Pharmacokinetics of Two Different Persantin® Sugar Coated Tablets in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 21.449
Record Dates: First submitted 2014-10-07; First posted 2014-10-09 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Healthy

ARMS (2):
- Persantin® new formulation (Experimental)
  Interventions: Drug: Persantin® new formulation
- Persantin® commercial formulation (Active Comparator)
  Interventions: Drug: Persantin® commercial formulation

INTERVENTIONS:
Drug: Persantin® new formulation
  Arms: Persantin® new formulation
Drug: Persantin® commercial formulation
  Arms: Persantin® commercial formulation

SUMMARY:
To investigate the relative bioavailability of the proposed formulation of PERSANTIN® compared to the present commercial formulation.

ELIGIBILITY:
Inclusion Criteria:

* All participants in the study should be healthy males, range from 21 to 50 years of age and their body mass index (BMI) be within 18.5 to 29.9 kg/m2
* All participants must give their written informed consent in accordance with Good Clinical Practice and local legislation prior to admission to the study

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug before enrolment in the study or during the study
* Use of any drugs which might influence the results of the trial up to 7 days prior to enrolment in the study or during the study
* Participation in another trial with an investigational drug (<= two months prior to administration or during the trial)
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation (>= 100 ml within four weeks prior to administration or during the trial)
* Any laboratory value outside the clinically accepted reference range
* Excessive physical activities within the last week before the trial or during the trial

Following exclusion criteria are of special interest for this study:

* History of haemorrhagic diathesis
* History of gastro-intestinal ulcer, perforation or bleeding
* Glucose-6-phosphate-dehydrogenase (G-6-PD) deficiency

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2001-10; Primary Completion 2001-12 (Actual)

PRIMARY OUTCOMES:
Area under the concentration time curve from 48 to 58 hours (AUC48-58) | 48 - 58 hours
Maximum concentration from 48 to 58 hours (Cmax48-58) | 48 - 58 hours

SECONDARY OUTCOMES:
Peak trough fluctuation (% PTF) | up to 48 hours
Minimum concentration from 48 to 58 hours (Cmin48-58) | 48 - 58 hours
Cmax48-58/AUC48-58 ratio | 48 - 58 hours
Time to maximum concentration from 48 to 58 hours (Tmax48-58) | up to 58 hours
Amount excreted in urine (Ae) | up to 24 hours after drug administration
Number of participants with adverse events | up to 8 days after last drug administration
Number of participants with clinically significant findings in vital functions | up to 8 days after last drug administration
  blood pressure, pulse rate
Number of participants with clinically significant findings in ECG | up to 8 days after last drug administration
Number of participants with clinically significant findings in laboratory tests | up to 8 days after last drug administration